CLINICAL TRIAL: NCT06270914
Title: Inclusive Positive Behavior Support in School - the Causal Mechanisms and Interactive Processes. A Study Protocol
Brief Title: Inclusive Positive Behaviour Supports
Acronym: IBIS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Principal Investigator, Martin Karlberg, Senior University Lecturer, Uppsala University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IBIS
Record Dates: First submitted 2024-01-27; First posted 2024-02-21 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Behavior Problem; Social Skills
Keywords: behavior problem; positive behavior support; prevention; universal
MeSH Terms: conditions — Mental Disorders; Social Skills | interventions — Palliative Care

STUDY DESIGN:
Intervention Model Description: This study utilizes quasi-experimental non-randomized design, including two waves of participant recruitment. Two waves of recruitment are used. In the first wave of recruitment, intervention and active control group are used and outcomes will be measured at three time points. In addition to quantitative data, qualitative observations and interviews are conducted to get a deeper understanding of the process of implementation of SWPIS. In the second wave of data recruitment, intervention and wait-list control group are used and outcomes will be measured at two time points (pre- and post).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Intervention (Experimental): The intervention group will receive the intervention Norwegian manualized program of SW-PBIS, N-PALS (Positiv Atferd, Støttende Læringsmiljø, og Sammhandling).
  Interventions: Behavioral: Inclusive Positive Behavior Interventions and Supports
- Active control (Active Comparator): Control group in the first wave of data collection is selected in accordance quasi-experimental design with nonequivalent control group. The teachers in the control group will, instead of a wait-list intervention, a shortened version of SW-PBIS containing only classroom leadership lectures. The schools that are part of the classroom management group also send staff for instructor training (ten training sessions, 25 hours in total, just as much as the SW-PBIS schools). Similar to the SW-PBIS group, the instructors in this group educate and supervise school staff, supported by a team at the school. Both groups have access to a manual and supporting materials. This design does not pose threats to the internal validity of the study, as classroom leadership is one of principles of PBIS framework. In this way it will be possible to explore the specific contribution of schoolwide PBS in contrast to classroom leadership only.
  Interventions: Behavioral: Inclusive Positive Behavior Interventions and Supports
- Control (No Intervention): Control group in the second wave of data collection constitutes a wait-list control group and will not be engaged in any kind of intervention during the intervention period.

INTERVENTIONS:
Behavioral: Inclusive Positive Behavior Interventions and Supports — The intervention is based on the Norwegian manualized program of SW-PBIS, N-PALS (Positiv Atferd, Støttende Læringsmiljø, og Sammhandling). The Norwegian model shares its core components with the original SW-PBIS model. The program's core components constitute: (a) positive behavior support strategies, including positive expectations and classroom rules, which are followed up with positive feedback and encouragement; (b) a system for monitoring student behavior, (c) school-wide corrections using consequences, (c) instruction in classroom management skills for teachers, and (e) strategies for collaboration with parents. These components are implemented through activities at school level and at classroom level.
  Arms: Active control; Intervention

SUMMARY:
Background: While positive school climate is important for students' well-being and mental health, school personnel may experience challenges in creating a nurturing school climate. School-Wide Positive Behavioral Interventions and Supports (SW-PBIS) have shown positive effects on school climate, but fewer studies have been conducted in the European context. Aim: The present project aims to investigate the effectiveness of SW-PBIS programs for students' social-emotional skills and academic achievement as well as teachers' and students' perceptions of the learning environment. Furthermore, the study intends to evaluate how school-level factors mediate or moderate the effects of the intervention. In addition, the study includes a qualitative evaluation of the dynamic interaction processes that occur during program implementation in local school contexts. Methods: Data on school- and individual-level measures are collected in intervention and control schools. With regard to challenges in retaining control groups over extended time periods, two waves of recruitment are used. In the first wave, an active control group is used, and data are collected during three time points. In the second wave, a wait-list control group is used, and data are collected during two time points during one school year. Hierarchical regression analyses will be conducted to explore the effects of SW-PBIS on the outcomes of the study. An ethnomethodological approach will be applied to provide a detailed examination of the social interactional and meaning-making practices of different school implementation teams, and the negotiation of normative expectations and rules of conduct in peer-teacher-student interactions in different classrooms. Discussion: The study is expected to contribute knowledge on the effects of the SWPBIS program and how these effects may be mediated or moderated by school-level factors. Combining quantitative and qualitative methods to explore the significance of school contexts in the implementation of the SWPBIS program constitutes the strength of the study. The challenge in the study is the extended period of implementation of SWPBIS, which entails difficulties in retaining a control group over the required time period. Therefore, two waves of recruitment are used, encompassing different procedures of allocation to intervention or control groups.

DETAILED DESCRIPTION:
Aim and Research Questions:

Firstly, the aim is to evaluate the effectiveness of the SWPBIS program for students' socio-emotional skills and academic achievement as well as teachers' and students' perceptions of the learning environment, and to explore how school-level factors may moderate or mediate the effect of SWPBIS on the outcomes. Secondly, the aim is to gain a deeper understanding of the social processes and local meanings that emerge and take form among the students, teachers, and other school professionals as they participate in the SW-PBIS program. The aims are specified in four research questions:

1. What are the effects of the SW-PBIS program on students' socio-emotional skills and academic achievement as well as teachers' and students' perceptions of the learning environment?
2. To what extent do school-level factors mediate and moderate the effects of the SW-PBIS program on the study outcomes over time?
3. How are the central contents of the SW-PBIS program made sense of and negotiated in school teams and classrooms at two schools during the course of program implementation?
4. How do specific instances of student-teacher interaction lead to changes in students' behavior and responses to the SW-PBIS program, and what forms of ethical dilemmas evolve in the management of behavior problems in classrooms?

Methods:

This study utilizes a quasi-experimental non-randomized design, including two waves of participant recruitment. In the first wave of recruitment, intervention and active control groups are used, and outcomes will be measured at three time points. In addition to quantitative data, qualitative observations and interviews are conducted to gain a deeper understanding of the process of implementing SWPIS. In the second wave of data recruitment, intervention and wait-list control groups are used, and outcomes will be measured at two time points (pre- and post).

The study will be conducted in compulsory schools and will include classes from grade four to grade nine. Each of the two waves of recruitment in the study will include 80 schools. Data will be collected on school-level measures and individual-level measures. School-level measures encompass: (a) Teacher collective self-efficacy; (b) Problem behavior in the classroom and school. Individual-level measures encompass: (a) Social-emotional skills; (b) Classroom environment; (c) Student achievement in national tests of mathematics and literacy.

The intervention is based on the Norwegian manualized program of SW-PBIS, N-PALS (Positiv Atferd, Støttende Læringsmiljø, og Samhandling). The Norwegian model shares its core components with the original SW-PBIS model. The program's core components constitute: (a) Positive behavior support strategies, including positive expectations and classroom rules, which are followed up with positive feedback and encouragement; (b) A system for monitoring student behavior, (c) School-wide corrections using consequences, (d) Instruction in classroom management skills for teachers, and (e) Strategies for collaboration with parents. These components are implemented through activities at the school level and at the classroom level. The implementation at the school level starts with establishing a leadership team, comprised of school leaders, team leaders, and members of the school welfare team. The leadership team assesses the needs and resources at the school and agrees on behavioral expectations and rules. The team monitors student behaviors and provides opportunities for teacher professional development with a focus on classroom management and relationship building. At the classroom level, the teachers incorporate school-wide expected behaviors into their classroom instruction through classroom activities and classroom rules. The teachers also integrate their training in classroom management and relationship building into their teaching practices. The duration of Tier 1 intervention is expected to be three years.

The control group in the first wave of data collection is selected in accordance with a quasi-experimental design with a nonequivalent control group. The teachers in the control group will, instead of a wait-list intervention, receive a shortened version of SW-PBIS containing only classroom leadership lectures. The schools that are part of the classroom management group also send staff for instructor training (ten training sessions, 25 hours in total, just as much as the SW-PBIS schools). Similar to the SW-PBIS group, the instructors in this group educate and supervise school staff, supported by a team at the school. Both groups have access to a manual and supporting materials. This design does not pose threats to the internal validity of the study, as classroom leadership is one of the principles of the PBIS framework. In this way, it will be possible to explore the specific contribution of schoolwide PBS in contrast to classroom leadership only. The control group in the second wave of data collection constitutes a wait-list control group and will not be engaged in any kind of intervention during the intervention period.

Hierarchical regression analyses with a three-level structure will be conducted to explore the effects of SW-PBIS on study outcomes. Hierarchical regression analyses allow for accounting for the nested structure of the data, in which teachers' and students' responses are nested within schools and grade levels. The outcomes at the school and individual levels will be studied as a function of time (three time points for wave 1 and two time points for wave 2) and group belonging (intervention or control group). To take into account the nestedness of the data, a three-level random effect model will be used, varying by school, grade, and the individuals' identification codes. Furthermore, the possible mediators (quality of implementation) and moderators (school characteristics, school-level variables) of the SWPBIS intervention will be analyzed. Missing data will be handled by imputation, provided that the assumption of data missing completely at random is met.

In the qualitative study, a longitudinal ethnographic approach will be used in order to obtain detailed contextualized knowledge on interactions in various contexts in two of the intervention schools, recruited in wave 1, over a longer period of time. Through purposeful sampling, three schools with different characteristics regarding size and catchment area will be selected.

ELIGIBILITY:
Inclusion Criteria:

* compulsory school, grades 4-9;
* the school have not been previously enrolled in an SWPBIS program by other providers;
* principal, teachers, students and their parents consent to participate in the study.

Exclusion Criteria:

* grades other than 4-9;
* the school has previously received or is enrolled in SWPBIS program or other PBS program;
* students or their parents have not consented to participation in the study.

Ages: 9 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 5000 (Estimated)
Dates: Start 2023-08-25 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Social emotional skills | 11 months
  Social Skills Improvement System - SEL Brief and Mental Health Scales, Teacher K-12 Form contains 20 items related to five competency domains (self-awareness, self-management, social awareness, relationship skills, and responsible decision making) and 10 items encompassing emotional behavior concerns (internalizing and externalizing concerns). Examples of items are "Asks for help when needed" for social-emotional skills competency domains and "Withdraws from others" for emotional behavior concerns. The items are measured on a 4-point scale (1=Never, 2=Seldom, 3=Often, 4=Almost always). The measures have proved to have sufficient validity and reliability in previous studies.
Classroom environment | 11 months
  A comprehensive assessment of the classroom learning environment was conducted using questionnaires for teachers and students. The teacher questionnaire consisted of 14 statements, rated on a 4-point scale (1 = does not fit to 4 = fits completely), assessing various aspects of the classroom learning climate. The student questionnaire included 22 statements, also rated on a 4-point scale, gauging students' perceptions of the classroom environment. An example of an item in the teacher questionnaire is "There is a good working climate during lessons". An example of an item in the student questionnaire is "Students in this class are active and interested during lessons".
Students' achievement | 11 months
  students' achievement on national tests of Swedish and mathematics will be retrieved from register data provided by Statistics Sweden. The data will be standardized across tests and compared with regard to the national average for those students who enter the project in grade 4 and 7 (national tests in grade 3 and grade 6) and finish the project in grade 6 and 9 (national tests in grade 6 and grade 9).

SECONDARY OUTCOMES:
Collective self-efficacy | 11 months
  Collective Self-efficacy questionnaire will be used as a measure of teacher collective beliefs of possibilities to influence student learning. CES contains 12 items and a 6-point scale is used (from 1=Do not agree at all, 2=Do not agree, 3=Do not agree fully, 4=Agree a little, 5=Agree, 6=Agree completely). An example of item is "Teachers in this school are able to get through to difficult students". In previous studies, collective self-efficacy has shown to be influenced by SWPBIS programs.
Problem behavior in classroom and school | 11 months
  Problem Behavior in the Classroom Last Week (20 items), in which the teachers are asked to report disruptive behavior on a 5-point Likert scale from 0 (not observed) to 5 (observed several times per day). Problem Behavior in the School Environment is a school level measure with similar structure and rating alternatives and is used with school staff. Examples of behaviors in the scales are "Destroying school environment" or "Physical aggression towards peers and teachers". The scales have shown satisfactory psychometric properties in several prior Norwegian studies.

OTHER OUTCOMES:
Implementation fidelity | 11 months
  To measure implementation fidelity of the SW-PBIS Tier 1, the members of school leadership team will be asked to complete questionnaire Benchmarks of Quality. The questionnaire is a self-evaluation tool that supports school professionals in monitoring progress of implementation of SW-PBIS Tier 1. BoQ contains 53 items, divided into 10 subscales covering team functioning, staff commitment, expectations and discipline procedures. Each item can be rated on a 3-point scale (1=Not yet, 2=Can be better, 3=Is in place). The items are summarized in a total score.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Education, Uppsala, Uppland, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Individual participant data will not be made available to other researchers due to ethical considerations.

REFERENCES:
- [Derived] Karlberg M, Klang N, Svahn J. Positive behavior support in school - a quasi-experimental mixed methods study and a randomized controlled trial. BMC Psychol. 2024 Oct 1;12(1):521. doi: 10.1186/s40359-024-02021-z. PMID 39354572